CLINICAL TRIAL: NCT01997671
Title: Effectiveness of an Intervention to Improve the Adequacy of the Indication of Lipid Lowering Treatment in Primary Prevention: Randomized Clinical Trial
Brief Title: Adequacy of the Indication of Lipid Lowering Treatment in Primary Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Preventive Services and Health Promotion Research Network (Other); Catalan Institute of Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EC11-342
Record Dates: First submitted 2013-01-25; First posted 2013-11-28 (Estimated); Last update posted 2013-12-02 (Estimated); Status verified 2013-11

CONDITIONS: Cardiovascular Diseases
Keywords: Primary Care; Lipid-lowering therapy; Prescription; Adequacy; Primary prevention; Cardiovascular diseases; Electronic Medical records; Clinical Practice Guideline
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Information Support System (Experimental): Practitioners in the intervention group may have access, whenever they want and through the computerized medical record program, to personalized information on their assigned patients who have started treatment of cardiovascular primary prevention with lipid-lowering.
  Interventions: Other: Information Support System
- Control group (No Intervention): Routine clinical practice

INTERVENTIONS:
Other: Information Support System — Practitioners in the intervention group may have access, whenever they want and through the computerized medical record program, to personalized information on their assigned patients who have started treatment of cardiovascular primary prevention with lipid-lowering. This information is updated monthly for 12 consecutive months.Information will be presented in two different and complementary ways to each practitioner: asynchronous information (the patient is not present when the practitioner receives the information) and synchronous information (the patient is present when the practitioner receives the information).
  Arms: Information Support System

SUMMARY:
OBJECTIVE: To evaluate the impact of an intervention addressed to health professionals to improve the adequacy of lipid-lowering prescription in primary prevention of cardiovascular disease and reducing expenditure in this respect.

DESIGN: a cluster randomized clinical trial, not blind; Data were obtained from medical records and other primary care databases.

SETTING: 279 primary health care teams in Catalonia (Spain), centers managed by Catalan Health Institute (ICS)

SUBJECTS: Population from 35 to 74 years, free of cardiovascular disease, who have been started on lipid-lowering therapy during 2 consecutive years of study.

INTERVENTION: Practitioners in the intervention group may have access, whenever they want and through the computerized medical record program, to personalized information on their assigned patients who have started treatment of cardiovascular primary prevention with lipid-lowering. This information is updated monthly for 12 consecutive months.Information will be presented in two different and complementary ways to each practitioner: asynchronous information (the patient is not present when the practitioner receives the information) and synchronous information (the patient is present when the practitioner receives the information).

VARIABLES:

1. Primary Outcomes are:

   * Variable RETIRA: new lipid-lowering treatments initiated during the year prior to the intervention, seen as inadequate and withdrawn during the intervention period.
   * Variable EVITA: New lipid-lowering treatments started during the intervention period and considered as inadequate.
2. Secondary Outcomes are:

   * Variable COST: total cost of the inadequate new lipid-lowering treatments.
   * Variable RECORD: recording of the cardiovascular risk.

2.Other variables:

* Principal: intervention/control group assignment of health professional.
* Patient variables: demographic and clinical.
* Professional variables: quality of care indicators.

STATISTICAL ANALYSIS: Descriptive analysis, agreggated at health professional level, will be performed and subsequently multilevel analysis techniques will be used to estimate the effect of intervention according to hierarchic data structure and, in particular, patient variables effect.

ELIGIBILITY:
Inclusion Criteria:

* Population from 35 to 74 years
* Free of cardiovascular disease
* Start on lipid-lowering therapy during 2 consecutive years of study

Exclusion Criteria:

* Previous treatment with lipid-lowering
* History of cardiovascular disease

Ages: 35 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60000 (Actual)
Dates: Start 2011-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
percentage of participants with increase of the adequacy of lipid-lowering prescription | up to 24 months
  The primary outcome is the improvement in the appropriateness of prescribing of lipid-lowering therapy in primary prevention as recommended by the guide clinical practice intervention in the Institut Català de la Salut compared with clinical practice group.
  To answer the main objective of the study, two dependent variables were calculated:
  * Variable RETIRA: new lipid-lowering treatments initiated during the year prior to the intervention, seen as inadequate and withdrawn during the intervention period
  * Variable EVITA: New lipid-lowering treatments started during the intervention period and considered as inadequate

SECONDARY OUTCOMES:
percentage of patients with cardiovascular risk register in the clinical records of patients | up to 24 months
  To assess the degree of cardiovascular risk register in the clinical records of patients RECORD variable is calculated:
  Variable RECORD: recording of the cardiovascular risk
Change from baseline in the total cost of the lipid-lowering treatments prescribed during the study period | baseline, months 24
  to assess the economic impact of the new primary prevention lipid-lowering treatments prescribed during the study period. To be determined by variable COST
  Variable COST: total cost of the inadequate new lipid-lowering treatments

CONTACTS AND LOCATIONS:
Overall Officials: Bonaventura Bolíbar, Principal Investigator — Jordi Gol i Gurina Foundation - IDIAP Jordi Gol; Sebastià Calero, Study Chair — Catalan Institute of Health; Josep Casajuana, Study Chair — Catalan Institute of Health; Ermengol Coma, Study Chair — Catalan Institute of Health; Francesc Fina, Study Chair — Catalan Institute of Health; Mireia Fàbregas, Study Chair — Catalan Institute of Health; Eduardo Hermosilla, Study Chair — Jordi Gol i Gurina Foundation - IDIAP Jordi Gol; Manolo Medina, Study Chair — Catalan Institute of Health; Mònica Monteagudo, Study Chair — Jordi Gol i Gurina Foundation - IDIAP Jordi Gol; Rosa Morros, Study Chair — Jordi Gol i Gurina Foundation - IDIAP Jordi Gol; Magdalena Rosell, Study Chair — Jordi Gol i Gurina Foundation - IDIAP Jordi Gol
Locations (1):
- IDIAP Jordi Gol, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Fabregas M, Berges I, Fina F, Hermosilla E, Coma E, Mendez L, Medina M, Calero S, Serrano E, Morros R, Monteagudo M, Bolibar B. Effectiveness of an intervention designed to optimize statins use: a primary prevention randomized clinical trial. BMC Fam Pract. 2014 Jul 15;15:135. doi: 10.1186/1471-2296-15-135. PMID 25027229